CLINICAL TRIAL: NCT04615546
Title: Role of Nutrient Transit and Incretin Hormones in Hyperinsulinemic Hypoglycemia
Brief Title: Role of Nutrient Transit in Hyperinsulinemic Hypoglycemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Tracey McLaughlin, Professor of Medicine, Endocrinology, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 52254
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Post-Bariatric Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Remote Phase: Post-Bariatric Hypoglycemia Patients (Experimental): Participants will wear continuous glucose monitor (CGM) in a blinded manner (cannot see data output) for 20 days followed by in an unblinded manner (can see data output) for 20 days.
  Interventions: Behavioral: Use of Continuous Glucose Monitor (CGM); Other: Use of "Cardea Solo" monitoring
- In-Clinic Phase: Post-Bariatric Hypoglycemia Patients (No Intervention): Participants will attend 1-3 study visits over the period of approximately 2 months, with metabolic parameters assessed under a variety of conditions. This group will also wear CGM during a portion of the metabolic tests. This may include participants from the Remote Phase or newly enrolled participants.
- In-Clinic Phase: Surgical Controls (No Intervention): Participants will attend 1-3 study visits over the period of approximately 2 months, with metabolic parameters assessed under a variety of conditions.
- In-Clinic Phase: Nonsurgical Controls (No Intervention): Participants will attend 1-3 study visits over the period of approximately 2 months, with metabolic parameters assessed under a variety of conditions.
- In-Clinic Phase: Post-Bariatric Hypoglycemia Patients with indwelling gastrostomy tube (No Intervention): Participants will undergo standardized mixed meal tolerance tests via oral, gastrostomy tube, and concomitant oral + gastrostomy tube routes of delivery with metabolic parameters assessed.

INTERVENTIONS:
Behavioral: Use of Continuous Glucose Monitor (CGM) — Participants will wear CGM
  Arms: Remote Phase: Post-Bariatric Hypoglycemia Patients
Other: Use of "Cardea Solo" monitoring — Participants will wear a "Cardea Solo" patch during blinded CGM use
  Arms: Remote Phase: Post-Bariatric Hypoglycemia Patients

SUMMARY:
Severe hypoglycemia (low blood sugar)after gastric bypass surgery is an increasingly recognized condition, characterized by symptoms of hypoglycemia after eating and inappropriately elevated insulin concentrations that occur at the time of hypoglycemia. Severe hypoglycemia can be dangerous and debilitating and can also impact cognitive function. At the moment no medical therapies have been developed for this disorder. Determining why some but not other patients develop this condition would allow for improved prediction, prevention, and treatment approaches. The purpose of the study is to understand the physiological changes observed in those patients who undergo gastric bypass and develop symptomatic hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18-70 years of age
* Post-bariatric surgery more than 6 months prior to signing the informed consent (not required for non-surgical controls)
* Documented history of hyperinsulinemic hypoglycemia (not required for post-bariatric and non-surgical controls)

Exclusion Criteria:

* Patients currently using sulfonylureas or other medications that may interfere with glucose metabolism within 5 half-lives of drug.
* Participation in any clinical investigation within 4 weeks prior to dosing
* History of or current insulinoma
* Active infection or significant acute illness within 2 weeks prior to dosing
* Female patients who are pregnant or lactating
* Women of childbearing potential and not utilizing effective contraceptive methods
* Inadequate end organ function as defined by: Serum creatinine >2.0 mg/dL, alanine transaminase (ALT) and aspartate aminotransferase (AST) > 2 x Upper Normal Limit
* Allergy to test meal or medications used in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-05-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Steady state plasma glucose (SSPG) as a measure of insulin sensitivity | Baseline 4-hour SSPG
  This endpoint applies to the In-Clinic Phase cohorts: Post-Bariatric Hypoglycemia, Surgical Controls, Non-Surgical Controls. This is a one day in-person appointment lasting approximately 6 hours.
Rate of gastric emptying | Baseline 4-hour scintigraphy procedure
  This endpoint applies to the In-Clinic Phase cohorts: Post-Bariatric Hypoglycemia, Surgical Controls, Non-Surgical Controls. This is an in-person appointment lasting approximately 5 hours.
Concentration of Glucagon-Like peptide 1 secretion augmentation of insulin secretion rate | Baseline 4-hour graded-glucose infusion
  This endpoint applies to the In-Clinic Phase cohorts: Post-Bariatric Hypoglycemia, Surgical Controls, Non-Surgical Controls. The blood collected from the SSPG will be stored and analyzed for the concentration of GLP-1 at multiple timepoints.
Rate of clinically important hypoglycemia (Level 2 hypoglycemia, <54 mg/dL) | 40 days
  This endpoint applies to Remote Phase participants
Percent time in clinically important hypoglycemia (Level 2 hypoglycemia, <54 mg/dL) | 40 days
  This endpoint applies to Remote Phase participants
Rate of arrhythmia during hypoglycemia | 10 days
  This endpoint applies to Remote Phase participants

CONTACTS AND LOCATIONS:
Overall Officials: Tracey McLaughlin, MD, Principal Investigator — Stanford University; Colleen Craig, MD, Study Director — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No